CLINICAL TRIAL: NCT00751478
Title: A Randomized, Double-Blind, Triple-Dummy, Single-Dose, Four-Way Crossover Study to Determine the Relative Bioavailability, Pharmacodynamic Effects, and Safety of Equivalent Doses of Whole and Crushed ALO-01 Versus Morphine IR in Opioid Experienced, Non-Dependent Subjects
Brief Title: Study to Determine the Bioavailability, Pharmacodynamic Effects, and Safety of Whole and Crushed ALO-01 Compared to Morphine Sulfate Immediate Release (MSIR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ALO-01-07-205
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: ALO-01; morphine; Determination of the relative pharmacodynamic effects; (including drug-liking), pharmacokinetics, and safety of; ALO-01 when administered whole or crushed and compared to; equivalent doses of immediate release morphine and placebo
MeSH Terms: conditions — Pressure Ulcer | interventions — morphine, naltrexone combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): 2 Placebo capsules (whole) + ALO-01 2 x 60 mg capsules (crushed) in apple juice + apple juice (MSIR placebo)
  Interventions: Drug: ALO-01
- B (Experimental): 2 x 60 mg ALO-01 (whole) + 2 x placebo capsules (crushed) in apple juice + apple juice (MSIR placebo)
  Interventions: Drug: ALO-01
- C (Active Comparator): 2 x placebo capsules (whole) + 2 X placebo capsules (crushed) in apple juice + 120 mg MSIR in apple juice
  Interventions: Drug: MSIR
- D (Placebo Comparator): 2 x placebo capsules (whole) + 2 X placebo capsules (crushed) in apple juice + apple juice (MSIR placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALO-01 — ALO-01 capsules
  Other Names: Morphine sulfate extended-release with sequestered naltrexone hydrochloride capsules
  Arms: A; B
Drug: MSIR — immediate release morphine sulfate
  Arms: C
Drug: Placebo — Placebo
  Arms: D

SUMMARY:
The purpose of the study is to determine the relative pharmacodynamic effects and safety of crushed and whole ALO-01 compared to MSIR and to Placebo, and of crushed ALO-01 to whole ALO-01; to determine the relative bioavailability of plasma morphine from crushed and whole ALO-01 compared to MSIR, and from crushed ALO-01 to whole ALO-01; and to determine the relative bioavailability of plasma naltrexone and 6-β-naltrexol from crushed ALO-01 to whole ALO-01.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 55 years of age, inclusive.
* Subjects had to be opioid users who were not currently physically dependent on opioids (based on DSM-IV criteria) but had experience in the use of opioids for non-therapeutic purposes (i.e. for psychoactive effects) on at least 10 occasions within last year and at least once in the 12 weeks prior to the screening session.
* Subjects had to be healthy as indicated by medical history, physical examination, vital signs, oxygen saturation, clinical laboratory tests, and 12-lead ECG performed at the screening session.
* Subjects had to consent to use two medically acceptable methods of contraception throughout the entire study period, including washout periods, and for females until one week after the study was completed.
* Female subjects had to have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the qualifying session and each treatment session, and not be lactating.
* Subject was willing and able to remain in the study unit for the entire duration of each confinement period and return to the study site for any outpatient visits.
* Subjects with a positive urine drug screen for opiates, amphetamines, cocaine and benzodiazepines at screening could enroll, provided they tested negative for the substances at the qualifying and each treatment session and had no clinically observed signs or symptoms of drug withdrawal.
* Subjects with a positive urine screen of tetrahydrocannabinol (THC) at screening could be enrolled, provided the THC levels were stable or decreasing on subsequent drug screens (prior to the qualifying and each treatment session).
* Subjects with body mass index (BMI) within the range 21-31 kg/m2 and weight greater than 55 kg, inclusive.
* Subjects had to voluntarily consent to participate in this study, provide their written informed consent prior to commencement of any study-specific procedures and understand that they were free to withdraw from the study at any time.

Exclusion Criteria:

Subjects excluded from the study were those:

* With a history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic or psychiatric disease or any other condition, which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
* With a history of clinically significant brain conditions (e.g., neoplasms, cerebrovascular disease, history of stroke, syncope, infectious disease or significant head trauma) or currently were being treated with medications or treatment regimens that lower seizure threshold.
* With a history or presence of drug or alcohol dependence excluding nicotine and caffeine. This included subjects who had ever been in a drug rehabilitation program.
* Who had a current psychiatric illness, except nicotine dependence. Subjects with a past history of psychiatric illness could be excluded at the discretion of the Investigator or designee.
* Who had a history of chronic obstructive pulmonary disease or any other lung disease (e.g., asthma) that could cause CO2 retention.
* Who had a clinically significant abnormal finding on the physical exam, medical history or clinical laboratory results at screening.
* Who had a history of allergic or adverse response to the study drugs or related drugs.
* Who had started a significantly restrictive diet during the four weeks preceding the first dose of study medication (qualifying session).
* Who had donated blood or plasma within 30 days prior to the first dose of study medication.
* Male subjects with hemoglobin less than 125 g/L and female subjects with hemoglobin less than 115 g/L.
* Who had participated in another clinical trial within 30 days prior to the first dose of study medication (qualifying session).
* Who had used any over-the-counter (OTC) medication, including vitamins and natural health products, within seven days prior to the first dose of study medication (qualifying session) without evaluation and approval by the study investigator.
* Who had used any prescription medication, except hormonal contraceptives or hormonal replacement therapy, within seven days prior to the first dose of study medication (qualifying session) without evaluation and approval by the study investigator.
* Who had a history of glaucoma or any other pupil abnormalities that in the opinion of the qualified investigator or designee could interfere with the ability to perform pupillometry.
* Who were not able to abstain from nicotine smoking while being in the clinical unit
* Who had had a positive test for or been treated for hepatitis B, hepatitis C or HIV.
* Who had current or pending legal charges.
* Who, in the opinion of the investigator, was not considered to be suitable and was unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pupillometry - Minimum Apparent Post-dose Pupil Diameter | Up to 24 hours post dosing
Pupillometry - Time to Minimum Apparent Post-dose Pupil Diameter | Up to 24 hours post dosing
VAS-Drug Liking - Peak effect (Emax) | Up to 24 hours post dosing
VAS-Drug Liking - Time of peak effect (TEmax) | Up to 24 hours post dosing
Cole/ARCI-Stimulation-Euphoria - Peak effect (Emax) | Up to 24 hours post dosing
Cole/ARCI-Stimulation-Euphoria - Time of peak effect (TEmax) | Up to 24 hours post dosing
VAS-High - Peak effect (Emax) | Up to 24 hours post dosing
VAS-High - Time of peak effect (TEmax) | Up to 24 hours post dosing

SECONDARY OUTCOMES:
Morphine Cmax | Up to 24 hours post dosing
Morphine Tmax | Up to 24 hours post dosing
Morphine AUC (0-8 h) | 0 - 8 hours post dosing
Morphine AUC (0-last) | Up to 24 hours post dosing
Morphine AUC (0-inf) | Up to 24 hours post dosing
Naltrexone Cmax | Up to 24 hours post dosing
Naltrexone Tmax | Up to 24 hours post dosing
Naltrexone AUC (0-8 h) | 0-8 hours post dosing
Naltrexone AUC (0-last) | Up to 24 hours post dosing
Naltrexone AUC (0-inf) | Up to 24 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Myroslav Romach, MSC, MD, Principal Investigator — DecisionLine Clinical research
Locations (1):
- DecisionLine Clinical Research, Toronto, Ontario, Canada